CLINICAL TRIAL: NCT02165943
Title: A Combined Retrospective and Prospective Protocol to Evaluate Vitoss With and Without Bone Marrow Aspirate for Benign Cavitary Lesions
Brief Title: Evaluation of Vitoss With and Without BMA for Benign Cavitary Lesions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Orthovita d/b/a Stryker (Industry)
Responsible Party: Sponsor
Other Study IDs: 1101-0014
Record Dates: First submitted 2014-05-30; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Bone Diseases
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitoss Bone Graft with BMA: Patients with a benign bone lesion of the extremity or pelvis for which surgical curettage age was recommended and who received Vitoss bone graft with BMA to fill the cavity.
  Interventions: Device: Vitoss
- Vitoss bone graft: Patients with a benign bone lesion of the extremity or pelvis for which surgical curettage was recommended and who received Vitoss bone graft to fill the cavity.
  Interventions: Device: Vitoss

INTERVENTIONS:
Device: Vitoss — Vitoss is a synthetic calcium-based bone void filler made of beta-tricalcium phosphate.

SUMMARY:
This is a retrospective, two-arm study reviewing the healing of cavitary defects in patients treated with Vitoss alone versus those treated with Vitoss with bone marrow aspirate (BMA). There will be a prospective follow-up visit at 24+ months to evaluate lont-term healing in patients identified during the retrospective portion of the study. It is thought that the inclusion of BMA will facilitate the resorption of the graft material, leading to better long-term bone healing.

ELIGIBILITY:
Inclusion Criteria:

* males and females >/= 18 years of age at the time of surgery
* Patients treated with Vitoss alone or Vitoss with added BMA between 2004 and 2012
* willing and able to provide Informed Consent to participate in and follow study requirements (including a radiologic assessment)

Exclusion Criteria:

* Patients with a known post-traumatic defect
* active infection at the time of implantation
* history of bone marrow disorders
* contraindications to the use of supplemental BMA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from retrospective records from the investigators specialty practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Vitoss resorption into the native bone as observed via CT | minimum of 24 months post-operatively
  Percentage of Vitoss resorption into the native bone will be retrospectively recorded in the Case Report Form at the 6 week, 3, 6, 12 and 18 month timepoints based on review of x-rays as well.

SECONDARY OUTCOMES:
Presence of graft within the soft tissue as observed by CT | minimum of 24 months post-operatively
  Presence of the graft within the soft tissue will be retrospectively recorded in the Case Report Form at the 6 week, 3, 6, 12 and 18 month timepoints based on review of x-rays as well.
Presence of a rim of radiolucency surrounding the grafted defect as observed by CT | minimum of 24 months post-operatively
  Presence of a rim of radiolucency surrounding the grafted defect will be retrospectively recorded in the Case Report Form at the 6 week, 3, 6, 12 and 18 month timepoints based on review of x-rays as well.
Size of the defect as observed by CT | minimum of 24 months post-operatively
  The size of the defect will be retrospectively recorded in the Case Report Form at the 6 week, 3, 6, 12 and 18 month timepoints based on review of x-rays as well.
Bone trabeculation through the defect as observed by CT | minimum of 24 months post-operatively
  Bone trabeculation through the defect will be retrospectively recorded in the Case Report Form at the 6 week, 3, 6, 12 and 18 month timepoints based on review of x-rays as well.
Persistence of graft material through the lesion as observed by CT | minimum of 24 months post-operatively
  Persistence of graft material through the lesion will be retrospectively recorded in the Case Report Form at the 6 week, 3, 6, 12 and 18 month timepoints based on review of x-rays as well.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Damron, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Upstate Orthopedics, LLC, Syracuse, New York, United States

REFERENCES:
- [Background] Bucholz RW, Carlton A, Holmes R. Interporous hydroxyapatite as a bone graft substitute in tibial plateau fractures. Clin Orthop Relat Res. 1989 Mar;(240):53-62. PMID 2537166
- [Background] Itokazu M, Matsunaga T, Ishii M, Kusakabe H, Wyni Y. Use of arthroscopy and interporous hydroxyapatite as a bone graft substitute in tibial plateau fractures. Arch Orthop Trauma Surg. 1996;115(1):45-8. doi: 10.1007/BF00453217. PMID 8775710
- [Background] Itokazu M, Matsunaga T. Arthroscopic restoration of depressed tibial plateau fractures using bone and hydroxyapatite grafts. Arthroscopy. 1993;9(1):103-8. doi: 10.1016/s0749-8063(05)80353-6. PMID 8442816
- [Background] McAndrew MP, Gorman PW, Lange TA. Tricalcium phosphate as a bone graft substitute in trauma: preliminary report. J Orthop Trauma. 1988;2(4):333-9. doi: 10.1097/00005131-198802040-00011. PMID 3074162
- [Background] Damron TA, Lisle J, Craig T, Wade M, Silbert W, Cohen H. Ultraporous beta-tricalcium phosphate alone or combined with bone marrow aspirate for benign cavitary lesions: comparison in a prospective randomized clinical trial. J Bone Joint Surg Am. 2013 Jan 16;95(2):158-66. doi: 10.2106/JBJS.K.00181. PMID 23324964
- [Background] Eggli PS, Muller W, Schenk RK. Porous hydroxyapatite and tricalcium phosphate cylinders with two different pore size ranges implanted in the cancellous bone of rabbits. A comparative histomorphometric and histologic study of bony ingrowth and implant substitution. Clin Orthop Relat Res. 1988 Jul;(232):127-38. PMID 2838207